CLINICAL TRIAL: NCT04906720
Title: Post-Ablation Pericarditis Reduction Study
Acronym: PAPERS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Vincent Cardiovascular Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R20200174
Record Dates: First submitted 2021-05-21; First posted 2021-05-28 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Atrial Fibrillation; Catheter Ablation; Pericarditis
MeSH Terms: conditions — Atrial Fibrillation; Pericarditis | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): Usual standard of care post atrial fibrillation ablation.
- Colchicine (Experimental): 0.6mg colchicine oral twice daily for 7 days.
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — colchicine 0.6mg oral twice daily for 7 days
  Other Names: colcrys; mitigare
  Arms: Colchicine

SUMMARY:
There has not been a prospective, randomized controlled trial of colchicine to reduce post-AF ablation pericarditis in an era of newer AF ablation techniques. The hypothesis is that an empiric pre and post AF ablation treatment protocol with colchicine may reduce the incidence and symptom severity of post-AF ablation related pericarditis. Thus, the goal of this study is to

1. Identify the incidence of post-AF ablation related pericarditis in patients undergoing ablation via high power, short duration strategy (shorter total RF time, but increased stability due to steerable catheters and possible difference from resistive vs conductive heating).
2. Identify potential differences in patients undergoing PVI only versus PVI + additional ablation
3. Identify whether patients on who are already on anti-inflammatories such as ASA or statins have a lower incidence than those without
4. Determine if an empiric treatment strategy with colchicine (for 7 days post ablation) reduces the incidence of post-operative AF

DETAILED DESCRIPTION:
This study will be a prospective, randomized controlled study of 248 patients presenting to the electrophysiology lab at Ascension St. Vincent (Indianapolis, IN) and Ascension Sacred Heart (Pensacola, FL) for atrial fibrillation ablation. Cases will be randomized in sequential order.

The control arm will undergo standard of care, whereas the study arm will undergo treatment with colchicine 0.6mg PO BID for 7 days following ablation.

Study variables will consist of

* Patient demographics

  o age, gender, comorbidities (HTN, HLD, DM-2, COPD, tobacco use, OSA, CKD, weight in kg, BMI, LVEF, autoimmune inflammatory condition such as RA), type of AF (paroxysmal, persistent, etc.)
* Medical therapy characteristics

  o anticoagulation choice, statin present, aspirin present, discontinuation of colchicine due to gastrointestinal distress
* Procedural characteristics o length of procedure, initial vs redo procedure, PVI only versus PVI + additional lines, total RF application time, HPSD vs MPMD approach, #RF applications, Power, Contact force, Impedance

Rates of acute post-operative pericarditis will be compared between the two groups. Subjects will be called by study personnel within 7-14 days to identify any post-ablation symptoms. If a patient develops pericarditis, standard anti-inflammatory therapy will be initiated in those patients regardless of study arm.

The primary outcome will be the development of post-AF ablation pericarditis within 30 days of ablation. This will be ascertained by comprehensive chart review and at the routine post-ablation follow up visit; additionally, there will be a standard telephone survey administered 7-14d after ablation (see instrument). Secondary outcomes will include symptoms, incidence of post-ablation AF recurrence, patient satisfaction using a Likert scale, and other clinical variables.

ELIGIBILITY:
Inclusion criteria:

- All patients >/= 18 undergoing atrial fibrillation ablation

Exclusion Criteria:

* Patients unable to receive or tolerate colchicine
* Pregnant or lactating women
* Concomitant use of drugs interacting with colchicine (including: cyclosporin, ranolazine, tacrolimus, clarithromycin, indinavir, itraconazole, ketoconazole, nefazadone, ritonavir, saquinavir, suboxone, telithromycin, erythromycin, fluconazole, verapamil, diltiazem, or more than 1 glass grapefruit juice daily)
* Severe renal impairment (CrCl < 30 mL/min)
* Severe hepatic impairment (ALT/AST greater than 5x ULN or clinical cirrhosis)
* Ongoing current use of colchicine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Pericarditis | Postoperative day 30.
  Clinical pericarditis ascertained by comprehensive chart review and a follow up phone call using a survey instrument.

SECONDARY OUTCOMES:
Proportion of patients with recurrent Atrial fibrillation | Through study completion, an average of 1 year
  Recurrence of atrial fibrillation post ablation
Median rating of patient satisfaction on a Likert scale, comparing the study group and standard of care group. | Postoperative day 14
  Patient satisfaction with ablation and post ablation care, measured on a Likert scale (min 1 and max 5, with 1 being best and 5 being worst) and derived from a telephone survey.

CONTACTS AND LOCATIONS:
Overall Officials: Parin J. Patel, MD, Principal Investigator — Physician; Board Member, Institutional Review Board; Board Member, Cardiovascular Research Institute
Locations (1):
- Ascension St Vincent Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leung YY, Yao Hui LL, Kraus VB. Colchicine--Update on mechanisms of action and therapeutic uses. Semin Arthritis Rheum. 2015 Dec;45(3):341-50. doi: 10.1016/j.semarthrit.2015.06.013. Epub 2015 Jun 26. PMID 26228647
- [Result] Imazio M, Bobbio M, Cecchi E, Demarie D, Demichelis B, Pomari F, Moratti M, Gaschino G, Giammaria M, Ghisio A, Belli R, Trinchero R. Colchicine in addition to conventional therapy for acute pericarditis: results of the COlchicine for acute PEricarditis (COPE) trial. Circulation. 2005 Sep 27;112(13):2012-6. doi: 10.1161/CIRCULATIONAHA.105.542738. PMID 16186437
- [Result] Imazio M, Brucato A, Ferrazzi P, Pullara A, Adler Y, Barosi A, Caforio AL, Cemin R, Chirillo F, Comoglio C, Cugola D, Cumetti D, Dyrda O, Ferrua S, Finkelstein Y, Flocco R, Gandino A, Hoit B, Innocente F, Maestroni S, Musumeci F, Oh J, Pergolini A, Polizzi V, Ristic A, Simon C, Spodick DH, Tarzia V, Trimboli S, Valenti A, Belli R, Gaita F; COPPS-2 Investigators. Colchicine for prevention of postpericardiotomy syndrome and postoperative atrial fibrillation: the COPPS-2 randomized clinical trial. JAMA. 2014 Sep 10;312(10):1016-23. doi: 10.1001/jama.2014.11026. PMID 25172965
- [Result] Tabbalat RA, Alhaddad I, Hammoudeh A, Khader YS, Khalaf HA, Obaidat M, Barakat J. Effect of Low-dose ColchiciNe on the InciDence of Atrial Fibrillation in Open Heart Surgery Patients: END-AF Low Dose Trial. J Int Med Res. 2020 Jul;48(7):300060520939832. doi: 10.1177/0300060520939832. PMID 32720823
- [Result] Deftereos S, Giannopoulos G, Kossyvakis C, Efremidis M, Panagopoulou V, Kaoukis A, Raisakis K, Bouras G, Angelidis C, Theodorakis A, Driva M, Doudoumis K, Pyrgakis V, Stefanadis C. Colchicine for prevention of early atrial fibrillation recurrence after pulmonary vein isolation: a randomized controlled study. J Am Coll Cardiol. 2012 Oct 30;60(18):1790-6. doi: 10.1016/j.jacc.2012.07.031. Epub 2012 Oct 3. PMID 23040570
- [Result] Deftereos S, Giannopoulos G, Efremidis M, Kossyvakis C, Katsivas A, Panagopoulou V, Papadimitriou C, Karageorgiou S, Doudoumis K, Raisakis K, Kaoukis A, Alexopoulos D, Manolis AS, Stefanadis C, Cleman MW. Colchicine for prevention of atrial fibrillation recurrence after pulmonary vein isolation: mid-term efficacy and effect on quality of life. Heart Rhythm. 2014 Apr;11(4):620-8. doi: 10.1016/j.hrthm.2014.02.002. Epub 2014 Feb 4. PMID 24508207
- [Result] Deyell MW, Leather RA, Macle L, Forman J, Khairy P, Zhang R, Ding L, Chakrabarti S, Yeung-Lai-Wah JA, Lane C, Novak PG, Sterns LD, Bennett MT, Laksman ZW, Sikkel MB, Andrade JG. Efficacy and Safety of Same-Day Discharge for Atrial Fibrillation Ablation. JACC Clin Electrophysiol. 2020 Jun;6(6):609-619. doi: 10.1016/j.jacep.2020.02.009. Epub 2020 Apr 29. PMID 32553209
- [Result] Ahmed AS, Clark BA, Joshi SA, Nair GV, Olson JA, Padanilam BJ, Patel PJ. Avoiding Bladder Catheters During Atrial Fibrillation Ablation. JACC Clin Electrophysiol. 2020 Feb;6(2):185-190. doi: 10.1016/j.jacep.2019.10.003. Epub 2019 Nov 27. PMID 32081221
- [Result] Gilge JL, Ahmed A, Clark BA, Slaten A, Devathu R, Olson JA, Padanilam BJ, Nair GV, Joshi SA, Ravichandran AK, Patel PJ. Left atrial hypertension and the risk of early incident heart failure after atrial fibrillation ablation. J Cardiovasc Electrophysiol. 2021 Feb;32(2):325-332. doi: 10.1111/jce.14829. Epub 2020 Dec 14. PMID 33270311